CLINICAL TRIAL: NCT00203840
Title: Pediatric Sleep Questionnaire: Normalization and Validation Study
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 13270A
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Sleep Disorders
Keywords: Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The information gathered from normal pediatric patients seen at the Pediatric Neurology Clinic in the DCAM and LaRabida Children's Hospital will be used to standardize and validate the information gathered from pediatric patients with sleep disorders. This will serve as the information source for a pediatric sleep database.

DETAILED DESCRIPTION:
A sleep questionnaire will be administered to patients who present to the Pediatric Neurology Clinic and LaRabida Children's Hospital. The questions asked are those routinely obtained in the clinical practice of sleep medicine. Medical students, residents and faculty as part of their normal clinical responsibilities will administer the questionnaire. The database will be maintained in Filemaker Pro program for future research purposes. Collection of the data will require approximately 15 minutes. A database file number not related to the patient medical record number will be assigned to each patient. The investigator will keep a separate log linking patient database number and patient medical record number. The logbook will be kept under lock and key by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen in the Pediatric Neurology Clinic and at LaRabida Children's Hospital

Exclusion Criteria:

* Adults

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: patients with sleep disorders
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2004-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pediatric Sleep Questionnaire | When data from clinic patients becomes available
  This questionnaire is used to better understand the natural history of sleeping disorders in children.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kohrman, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States